CLINICAL TRIAL: NCT03885193
Title: Impact of HMS Plus Device on Postoperative Blood Loss During Cardiac Surgery
Acronym: POC/HMS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0063
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Surgical Procedure
Keywords: anticoagulation; cardiopulmonary bypass; heparin; protamine; postoperatively bleeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HMS plus group: HMS plus device is employed to assess anticoagulation and ensure adequate heparin and protamine dosing during cardiopulmonary bypass (CPB).
- ACT plus group: ACT plus device is employed to assess anticoagulation and ensure adequate heparin and protamine dosing during cardiopulmonary bypass (CPB).

SUMMARY:
Activated clotting times (ACT) is employed most commonly to assess anticoagulation and ensure adequate heparin and protamine dosing during cardiopulmonary bypass (CPB). However, many studies have demonstrated a lack of correlation between plasma heparin levels and ACT during CPB.

HMS Plus device estimate the free plasma heparin level from a whole-blood sample and also include the dose of protamine necessary to neutralize the circulating heparin at the end of CPB. It could predict a higher heparin dose and lower protamine dose but it's interest on postoperative bleeding and perioperative transfusion is unclear.

DETAILED DESCRIPTION:
Adult cardiac surgery is often complicated by elevated blood losses that account for elevated transfusion requirements. Perioperative bleeding and transfusion of blood products are major risk factors for morbidity and mortality.

Cardiac surgery is a challenge in the management of coagulation because of the requirement for both a fully anticoagulated state for CPB and a return-to-normal hemostasis at its conclusion. Conditions during CPB, such as hemodilution, hypothermia, platelet activation and coagulopathy are know to cause falsify elevated ACT readings. For these reasons, relying on the ACT alone may lead to inadequate anticoagulation.

Moreover, no consensus about the monitoring or level of anticoagulation required has been reached. Similarly, the neutralization of heparin is performed with protamine (dose/dose). This empirical approach does not include inter- and intra-individual variations, which can involve bleeding complications. By using the HMS Plus, heparin and protamine dosing are individualized based on each patient's responsiveness to heparin, eliminating the need for empiric weight-based dosing.

HMS Plus provided a rapid assessment of heparin concentration that correlated well with anti-Xa assays. This could attenuates this hemostatic activation by decreasing excessive generation of thrombin and plasmin. Also, this ensures preservation of coagulation factors and decreases thrombin-mediated consumption and activation of platelets during CPB.

HMS Plus is ability to calculate the amount of circulating heparin at the end of CPB and give the exact dose of protamine necessary to neutralize the heparin. Targeted dosing can prevent excessive protamine administration and reduce protamine-induced platelet dysfunction.

In a meta-analysis of 4 randomized controlled trials involving a total of 507 patients, postoperatively blood loss was lower in the HMS group compared with the control group. But the supporting studies were limited by small sample sizes, outdated practice techniques, not involve surgery at risk and have liberal transfusion practices. Moreover, studies observed errors in calculating the heparin bolus dose with HMS Plus if patient had an inadequate antithrombin level. The administration of more heparin is a cause of heparin rebound in the postoperative period and potentially was increasing the risk for bleeding.

So, it would be necessary to compare ACT Plus and HMS Plus devices on postoperatively bleeding in a study involve patients at risk to bleeding and with a transfusion protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with cardiopulmonary bypass (valve procedure, coronary artery bypass grafting (CABG), heart transplantation,..)

Exclusion Criteria:

* Minors
* Isolated aortic valve procedure unless high risk of hemorrhage (endocarditis, redo surgery)
* Contra indication to heparin and/or protamine

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery with cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
postoperative bleeding in cardiac surgery | First 24 hours
  Compare HMS Plus and ACT Plus devices on postoperative bleeding in cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France